CLINICAL TRIAL: NCT03730090
Title: Hypothermia in Cesarean Sectio Patients in Regional Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Other Study IDs: Hypothermia Sectio OUS
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: zero flux skin termometer — Core temperature is monitored continously, non-invasively

SUMMARY:
To study the core temperature perioperatively in patients due for elective cesarean sectio in spinal anaesthesia.

Core temperature will be registered by a zero-flux (SpotOn. 3m) probe on the forehead, starting in the holding area and continued until normotemperature post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients
* planned spinal anaesthesia

Exclusion Criteria:

* Conversion of procedure to general anaesthesia
* allergy to temperature probe (adhesive)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female patients for sectio
Study Population: consecutive, elective cesarean sectio
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
incidence of perioperative hypothermia, less than 36.0 degrees | perioperatively
  mesured by zero flux in forehead

SECONDARY OUTCOMES:
patient satisfaction: Patient will be asked to grade | perioperatively, repeated
  Patient will be asked to grade their feeling of being Cold/warm
duration of perioperative hypothermia | perioperatively, continously
  number of minutes below 36.0 degrees
shivering | perioperatively
  any shivering due to being cold

IPD SHARING:
Plan to Share IPD: Undecided